CLINICAL TRIAL: NCT07399301
Title: Effect of High-Intensity Functional Training on Physical Performance and Mental Health in Elderly With Sarcopenia
Brief Title: High-Intensity Functional Training on Physical Performance and Mental Health in Elderly With Sarcopenia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Neveen Mohammed Ibrahim Nawar, Physiotherapy Specialist at Damanhur Medical National Institute, EL-Behira, Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202663
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Geriatric Sarcopenia
Keywords: HIGH- INTENSITY FUNCTIONAL TRAINING- PHYSICAL PERFORMANCE - MENTAL HEALTH - ELDERLY - SARCOPENIA
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high-intensity functional training exercises (Experimental): A) Awarm up: for 5 min, B) Functional training exercises: The participants will be initially instructed to complete up to one set of 8 maximum repetitions for each type of exercise with first and second week, followed by two sets of 8 maximum repetitions in the third and fourth week, Then three sets of 12 maximum repetitions from the fifth week untile the end of the study I. Sit to stand( Chair squats)
  II. Wall push up:
  III. Overhead triceps extension:
  IV. Leg kickbacks V. Wood chops exercise VI. Farmer's Carry training C) A cool down: for 5 min slow continuation of the activity.
  Interventions: Other: High-Intenisity Functional Training
- sham therapy (Sham Comparator): Group (B): N=30 Patients in this group who will be found to have sarcopenia will receive sham exercises. Sham interventions are methodological tools used to treat participants in the study arm and the control arm in exactly the same way, except that the study group receives an active substance and the control group does not.Sham exercises that is commonly administrated as a light touch in the body or mimics the active treatment and aims at blinding of participants
  Interventions: Other: Sham

INTERVENTIONS:
Other: High-Intenisity Functional Training — A) Awarm up: for 5 min.warm-up (predominantly stretching) of the neck, shoulders, lower back, hips, knees and ankles.
  B) Functional training exercises: The participants will be initially instructed to complete up to one set of 8 maximum repetitions for each type of exercise with first and second week, followed by two sets of 8 maximum repetitions in the third and fourth week, Then three sets of 12 maximum repetitions from the fifth week untile the end of the study.
  I. Sit to stand( Chair squats) II. Wall push up III. Overhead triceps extension IV. Leg kickbacks V. Wood chops exercise VI. Farmer's Carry training C) A cool down: for 5 min slow continuation of the activity, allows a more gradual reduction in heart rate and increased peripheral vascular resistance, with return of blood flow from the periphery Farmer's Carry training
  Arms: high-intensity functional training exercises
Other: Sham — The participants in the control group will receive sham exercises that is commonly administrated as a light touch in the body or mimics the active treatment and aims at blinding of participants.
  Arms: sham therapy

SUMMARY:
Sixty patients with age ranged from 60 to 70 years old with individuals who will be found to have sarcopenia will participate in the study, and will be recruited from nursing home in AL-Abadiyah.

Patients will be assigned into two equal groups randomly:

Group(A):N= 30

Patients in this group will receive high-intensity functional training exercises 3 times per week for 10 weeks. The initial duration of each session was 30 min, and it could be increased progressively, along with the intensity of the exercises, up to 50 min. All sessions included the following:

i. 5 min warm-up ii. 40 min functional training exercises. iii. 5 min cool-down. Group (B): N=30 Patients in this group will receive sham exercises. Sham interventions are methodological tools used to treat participants in the study arm and the control arm in exactly the same way, except that the study group receives an active substance and the control group does not.

DETAILED DESCRIPTION:
Sixty patients with age ranged from 60 to 70 years old with individuals who will be found to have sarcopenia will participate in the study, and will be recruited from nursing home in AL-Abadiyah.

Patients will be assigned into two equal groups randomly:

Group (B): N=30 Patients in this group will receive sham exercises. Sham interventions are methodological tools used to treat participants in the study arm and the control arm in exactly the same way, except that the study group receives an active substance and the control group does not.The participants in the control group will receive sham exercises that is commonly administrated as a light touch in the body or mimics the active treatment and aims at blinding of participants

Procedures:

(A)Evaluating procedures: Before starting the exercise program, a complete history and physical examination will be taken from each subject. Each subject of the two groups will undergo the following steps of measurements. The parameters will be recorded at the beginning and the end of the total study period (10 weeks).

1. Hand Dynamometer.
2. Short Physical Performance.
3. Quadriceps strength test
4. Montreal Cognitive Assessment
5. The Katz Index.
6. The Geriatric Depression Scale-15 (GDS-15).
7. The UCLA Loneliness Scale (Version 3). (B) Intervention procedures: All patients will be classified into two equal groups; each group will consist of 30 patients.

I-Intervention for Group A :

Patients in this group will receive high-intensity functional training exercises 3 times per week for 10 weeks. The initial duration of each session was 30 min, and it could be increased progressively, along with the intensity of the exercises, up to 50 min. All sessions included the following:

i. 5 min warm-up ii. 40 min functional training exercises. Functional training exercises: The participants will be initially instructed to complete up to one set of 8 maximum repetitions for each type of exercise with first and second week, followed by two sets of 8 maximum repetitions in the third and fourth week, Then three sets of 12 maximum repetitions from the fifth week untile the end of the study.

I. Sit to stand( Chair squats) II. Wall push up III. Overhead triceps extension IV. Leg kickbacks V. Wood chops exercise VI. Farmer's Carry training C) A cool down: for 5 min

II. Intervention for Group B :

The participants in the control group will receive sham exercises that is commonly administrated as a light touch in the body or mimics the active treatment and aims at blinding of participants.

ELIGIBILITY:
Inclusion Criteria: INCLUSION CRITERIA:

1. Old individuals who will be found to have sarcopenia as defined according to European Working Group on Sarcopenia in Older People (EWGSOP2) 2019 criteria, The EWGSOP2 defines sarcopenia as a muscle disease characterized by progressive and generalized loss of skeletal muscle mass and function. Diagnosis requires sequential assessment of three components

   * Low Muscle Strength: The primary criterion. Measured by:

     * Handgrip strength: Cut-offs are <27 kg for men and <16 kg for women using a dynamometer.
     * Chair Stand Test: ≥15 seconds for five rises indicates weakness.
   * Low Muscle Quantity or Quality: Assessed via:

     o calf circumference (≤34 cm men, ≤33 cm women).
   * Poor Physical Performance: Indicates severe sarcopenia. Tests include:

     * Gait speed: ≤0.8 m/s over 4 meters.
     * Short Physical Performance Battery (SPPB): ≤8 points.
     * Timed Up-and-Go (TUG): ≥20 seconds.
2. Age from 60 to 70 years old.
3. Old individuals who will be found to have mild depression.

Exclusion Criteria:

1. Neurological disorders.
2. Vestibular or balance disorders.
3. Uncontrolled hypertension or heart diseases.
4. Recent surgeries or fractures.
5. Any psychological disorders.
6. Severe renal failure (glomerular filtration rate < 30 mL/min).
7. moderate to severe liver failure.
8. The patients cannot follow instructions.

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) test | 10 weeks
  The SPPB assesses physical performance through balance, strength, and gait measurements and is made up of a set of three tests: standing static balance ; lower limb strength and power through getting up and sitting on a chair; and walking speed at normal pace. Strength and gait are first evaluated by the ability to perform the tasks of getting up and sitting on a chair five times and performing the walking speed test (3 to 4 meters) and, second, by the time the individual takes to complete the tasks. The SPPB total score ranges from 0 (worst performance) to 12 points (best performance) and categorically evaluates performance in the tests using three classes of scores: three classes: 0-6 points (poor performance), 7-9 points (moderate performance), and 10-12 points (good performance).

SECONDARY OUTCOMES:
Hand Dynamometer | 10 weeks
  Are portable devices usually incorporating a wireless load cell with an inbuilt microprocessor to measure isometric muscle force across both clinical and healthy populations.To assess hand grip, participants will sit in a chair with their feet support. The hand and forearm will assess by position with the shoulder adducted and in neutral rotation, with the elbow in 90◦ of flexion, forearm in neutral, and the wrist in 0 to 30◦ of extension and 0 to 15◦ of ulnar deviation. The participant will ask to grasp the hand-held dynamometer with the fingers wrapped around the handle. The clinical evaluator instructed the participant to perform a maximal contraction lasting three to five seconds, saying, "when I say go, I want you to squeeze the handle as hard as you can.
Quadriceps strength test | 10 weeks
  manual muscle testing (MMT) is a highly reliable method for assessing strength. The patient is sitting upright and positioned to allow full movement of the joint against gravity. The examiner will demonstrate the desired movement against gravity. Verbal instructions; "Straighten your knee". The hand will give resistance on top of the leg just proximal to the ankle. The other hand is placed under the thigh above the knee.
Montreal Cognitive Assessment | 10 weeks
  Is a diagnostic test for Mild cognitive impairment. A score of 90 or more indicates normality, 89-78 is an indication of MCI, and a score lower than 78 is diagnostic for dementia.
The Katz Index | 10 weeks
  Is designed to assess functional status, specifically, the individual's ability to perform activities of daily living (ADLs) independently. The index ranks the performance in the following six functions: bathing, dressing, toileting, transferring, continence, and feeding. If no supervision, direction, or personal assistance is required, then 1 point is given to that functional activity. If the individual requires supervision, direction, personal assistance, or total care, then a 0 is assigned to that functional activity. A total score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less indicates severe functional impairment.
The Geriatric Depression Scale-15 (GDS-15) | 10 weeks
  The scale contains 15 items, and the answers are composed of "yes/no", with the total score ranging from 0 to 15. The scale mainly evaluates the depression status of participants in the recent week.The total score >5 was classified as depression positive
The UCLA Loneliness Scale (Version 3) | 10 weeks
  the measure was highly reliable, both in terms of internal consistency and test-retest reliability over a 1-year period. Hardly ever or never = 1; some of the time = 2; often = 3. The lowest possible combined score on the loneliness scale is 3 (indicating less frequent loneliness) and the highest is 9 (indicating more frequent loneliness)

CONTACTS AND LOCATIONS:
Overall Officials: Research Ethical Committee Faculty of Physical Therapy - Cairo University, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt